CLINICAL TRIAL: NCT05283850
Title: A Prospective, Pre-Hospital Comparison of Normal Saline Versus Half-Normal Saline, After Universal Calcium Chloride Administration, to Improve Outcomes in Pulseless Electrical Activity Patients
Brief Title: Surviving PEA in Roanoke (SPEAR) Study
Acronym: SPEAR
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Carol Bernier (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor-Investigator, Carol Bernier, Assistant Professor of Emergency Medicine, Carilion Clinic
Organization: Carilion Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-19-488
Record Dates: First submitted 2022-02-20; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Cardiac Arrest; Pulseless Electrical Activity
Keywords: Crystalloid Fluids; Emergency Medical Services (EMS); Pre-Hospital Medicine; Sodium Chloride; Calcium Chloride; Normal Saline; Half-Normal Saline; Waiver of Informed Consent; Paramedic; Electrolyte
MeSH Terms: conditions — Heart Arrest | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, being intrinsically unconscious from PEA, will be blinded to the intervention. EMS Supervisors, in the pre-hospital setting, will administer an opaque bag of fluids with only a bag number on it, ensuring that they are blinded to the intervention. Hospital providers/outcomes assessors will know that patients were enrolled in a study and they will only know which bag number was used. The investigator will have the capacity to unblind bag numbers, but the investigator will not be the provider or outcomes assessor for patients due to the emergent nature of PEA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High-Calcium, High- Sodium (HCHS) group (Active Comparator): Patients will receive a drip of blinded, intravenous, normal saline and an unblinded, intravenous, one gram bolus of calcium chloride.
  Interventions: Drug: High Calcium, High Sodium (HCHS) Crystalloid Therapy
- High-Calcium, Low- Sodium (HCLS) group (Experimental): Patients will receive a drip of blinded, intravenous, half-normal saline and an unblinded, intravenous, one gram bolus of calcium chloride.
  Interventions: Drug: High Calcium, Low Sodium (HCLS) Crystalloid Therapy

INTERVENTIONS:
Drug: High Calcium, Low Sodium (HCLS) Crystalloid Therapy — Half-normal saline IV drip and 1g IV bolus Calcium Chloride.
  Other Names: (NDC) National Drug Code NDC 0264-7800-00 and NDC 0409-4928-11
  Arms: High-Calcium, Low- Sodium (HCLS) group
Drug: High Calcium, High Sodium (HCHS) Crystalloid Therapy — Normal saline IV drip and 1g IV bolus Calcium Chloride.
  Other Names: NDC NDC 0264-7802-00 and NDC 0409-4928-11
  Arms: High-Calcium, High- Sodium (HCHS) group

SUMMARY:
The Carilion Clinic and Virginia Tech Carilion School of Medicine, in conjunction with Roanoke Fire-EMS, Botetourt County Department of Fire & EMS and Salem Fire-EMS, are studying the outcomes of patients experiencing Pulseless Electrical Activity (PEA). PEA refers to a type of cardiac arrest in which there is normal electrical activity in the heart however the heart still fails to contract to generate a pulse. Without heart contractions, which normally generates a pulse, the brain and other important organs fail to receive blood and oxygen. Unfortunately, the majority (97.3%) of patients that experience this rhythm do not survive and most don't even make it to the hospital. This study is trying to determine if the administration of a High Calcium, Low Sodium (HCLS) fluid in pre-hospital care will improve the chances of survival.

Generally, a sodium (salt) solution is provided to patients experiencing cardiac arrest. Studies have shown that lower sodium and higher calcium content may activate certain parts of the heart cells required to generate a pulse under PEA conditions.

This study is a double-blind, prospective, clinical trial. PEA patients will randomly receive either routine fluid therapy (salt solution) or a HCLS solution. While HCLS solution is not the standard fluid used by EMS providers responding to PEA, it is composed of FDA approved components and is occasionally used by EMS providers at their discretion in treating PEA. It is predicted that HCLS will either improve PEA survival or deliver similar outcomes as routine treatment. All patients will receive standard, high quality cardiac arrest and post-cardiac arrest care regardless of assigned treatment group.

DETAILED DESCRIPTION:
Pursuant to a Waiver of Informed Consent, this investigation will automatically enroll all eligible PEA patients treated by Roanoke Fire-EMS, Botetourt County Department of Fire & EMS and/or Salem Fire-EMS systems.

Once patients are enrolled, they will be de-facto randomized into one of two groups: control High Calcium-High Sodium (HCHS) or interventional High Calcium-Low Sodium (HCLS). Supervisors will have on their trucks, numbered-but-otherwise-blinded bags of half-normal saline or normal saline solution. The bags will be numbered, recorded and randomized by this study's investigators. Supervisors, when providing care, will universally administer 1g unblinded CaCl2 and then subsequently chose a crystalloid fluid set to use from their trucks randomly. The crystalloid will be administered as a wide open IV drip at a rate of at least 1000ml/hour, depending on gauge size, for as long as fluids are indicated for, likely resulting in a crystalloid dose of 0.5-2(L) liters. Each bag-set will have two bags of the same blinded unit to allow for treatment with up to (2L) 2 liters of fluid for a patient. Explicitly, all enrolled patients will be receiving calcium, it is only the crystalloid fluid (normal saline vs half-normal saline) that will differ. HCLS treatment was designed to be hyponatremic compared to normal saline (while both groups in this trial will be hypercalcemic compared to pure normal saline PEA therapy) in order to initiate low sodium inotropy.

The contents of the bag will be blinded to the supervisor. Neither the patient nor the supervisor will know which treatment was given thus ensuring double-blinding. Further, by randomly choosing a bag with no knowledge of its contents, the treatment will effectively be randomized. Both groups will otherwise receive current routine Advanced Cardiac Life Support and either standard post-arrest care or standard termination of care. Per Roanoke Fire-EMS, Botetourt County Department of Fire & EMS and Salem Fire-EMS standard protocol, only patients who undergo ROSC on scene will be transported to a hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients who present with PEA at any time during the patients' treatment by Roanoke Fire-EMS, Botetourt County Department of Fire & EMS and/or Salem Fire-EMS. This study defines a PEA presentation as any patient who is unconscious, presenting without a carotid pulse and with non-(VT/VF) ventricular tachycardia/ventricular fibrillation electrical activity.

Exclusion Criteria:

* Patient less than 18 years old
* Known pregnancy
* Duration of untreated cardiac arrest of more than 30 minutes
* Traumatic cardiac arrest
* Known (LVAD) Left Ventricular Assist Device
* Rapidly fatal underlying disease
* Known or suspected digitalis toxicity
* A physical, durable (DNR) Do Not Resuscitate (or durable DNR medical jewelry) presented to EMS before treatment with asserting a preference not to be enrolled
* Prisoners and other populations with involuntary consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Event Survival | Up to 1 hour
  ROSC sustained until arrival at the emergency department and transfer of care to medical staff at the receiving hospital?

SECONDARY OUTCOMES:
Any Return-Of-Spontaneous-Circulation (ROSC) | Through resuscitation efforts up to 1 hour after arrival to (ED) Emergency Department
  Did the patient achieve ROSC at any point during the resuscitation attempt?
Survival to hospital discharge | Up to 30 days after admission to (ED) Emergency Department
  Did the patient survive to hospital discharge?
Neurological outcome at hospital discharge | Up to 30 days after admission to ED
  (CPC) Cerebral Performance Category Score and/or (mRS) modified Rankin Score at hospital discharge?
Serum Electrolyte Values | Up to 12 hour after admission to the (ED) Emergency Department
  All (BMP) Basic Metabolic Panel values will be collected, but there is a particular emphasis on serum sodium and calcium values.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Bernier, DO, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Unidentified data could be arranged to be shared with researchers who specifically request it, but this study is not currently (IRB) Institutional Review Board approved to do so.